CLINICAL TRIAL: NCT00005485
Title: The Jackson Heart Study of Cardiovascular Disease Among African Americans
Acronym: JHS
Status: Active, not recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 5001; HHSN268201800010I (Other Grant/Funding Number: NHLBI and NIMHD); HHSN268201800011I (Other Grant/Funding Number: NHLBI and NIMHD); HHSN268201800012I (Other Grant/Funding Number: NHLBI and NIMHD); HHSN268201800013I (Other Grant/Funding Number: NHLBI and NIMHD); HHSN268201800014I (Other Grant/Funding Number: NHLBI and NIMHD); HHSN268201800015I (Other Grant/Funding Number: NHLBI and NIMHD)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Disease; Hypertension; Cerebrovascular Disorders
Keywords: Cardiovascular diseases; Heart failure; Stroke; Coronary heart disease; Diabetes; Hypertension; Chronic kidney disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Disease; Hypertension; Cerebrovascular Disorders; Heart Failure; Stroke; Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, urine, DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective study of the environmental and genetic factors that influence the development of cardiovascular disease (CVD) in African American adults. The cohort is a collaboration among multiple institutions (Jackson State University, Mississippi State Department of Health, Tougaloo College, and the University of Mississippi Medical Center), NIMHD, and NHLBI.

DETAILED DESCRIPTION:
The Jackson Heart Study (JHS) initiated in 1998, is a longitudinal investigation of genetic and environmental risk factors associated with the disproportionate burden of cardiovascular disease (CVD) in African American adults. In addition, the JHS conducts community education and outreach activities to promote healthy lifestyles and reduce disease risk burden, undergraduate- and graduate-level research training programs, and high school science and math enrichment programs to prepare and encourage students to pursue biomedical careers. The study recruited 5306 African American adults living in the Jackson, MS area (Hinds, Madison, and Rankin Counties). Participants were enrolled from each of 4 recruitment pools: random, 17%; volunteer, 30%; currently enrolled in the Atherosclerosis Risk in Communities (ARIC) Study, 31% (shared JHS/ARIC cohort); and secondary family members, 22%. Recruitment was limited to non-institutionalized African American adults aged 35-84 years, except in a nested family cohort where those aged 21+ years were also eligible. Among those enrolled, approximately 3,700 gave consent that allows genetic research and deposition of data into dbGaP. JHS participants have completed four clinical examinations (Exam 1, 2000-04; Exam 2, 2005-08; Exam 3, 2009-13; Exam 4, 2021-2025) that have generated extensive longitudinal data on traditional and putative CVD risk factors, socioeconomic and sociocultural factors, biochemical analytes, and measures of subclinical disease from echocardiography, cardiac magnetic resonance imaging (MRI), and computed tomography (CT) scans of the heart, aorta, and abdomen. Stored biological samples have been assayed for putative biochemical risk factors and stored for future research. DNA has been extracted and lymphocytes cryopreserved for study of candidate genes, genome-wide scanning, expression, and other -omics investigations. Participants have been contacted annually to update information, confirm vital status, document interim medical events, hospitalizations, and functional status, and obtain additional sociocultural information. Ongoing cohort surveillance includes abstraction of medical records and death certificates for relevant International Classification of Diseases (ICD) codes and adjudication of nonfatal events and deaths. The JHS serves as a resource to the scientific community for novel research, promotes cardiovascular health in the local community, and encourages students and fellows to pursue biomedical careers.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Residents of Jackson, Mississippi

Exclusion Criteria:

* Institutionalization

Ages: 35 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African-American adult residents of metropolitan Jackson, Mississippi
Sampling Method: Non-Probability Sample
Enrollment: 5306 (Actual)
Dates: Start 2000-09-19 (Actual); Primary Completion 2025-08-12 (Estimated); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Disease | 2000-2016
  Coronary Heart Disease, Stroke, Heart Failure

SECONDARY OUTCOMES:
Mortality | 2000-2018
  All Cause

CONTACTS AND LOCATIONS:
Overall Officials: Wendy White, PhD, Principal Investigator — Tougaloo College JHS UTEC; Marinelle Payton, MD, PhD, Principal Investigator — Jackson State University JHS GTEC; April P Carson, PhD, Principal Investigator — UMMC JHS CC and FC; Victor Sutton, PhD, Principal Investigator — Mississippi State Department of Health JHS CEC; Jennifer Reneker, PhD, Principal Investigator — UMMC JHS GTEC
Locations (1):
- UMMC, JSU, Tougaloo College, MSDH, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
The JHS adheres to NIH and NHLBI policies for data sharing of epidemiologic studies. Data from each cycle of an examination or follow-up component are prepared by the JHS Coordinating Center and sent to the NHLBI PO for distribution as a data set after the completion of each examination or two years after the baseline, follow-up, genetic, ancillary study, or other data set is finalized within the study for analysis for use in publication. De-identified data from Exams 1, 2 and 3 of the JHS are available and shared commonly through the JHS processes for presentation and publication and ancillary studies. Public datasets for Exam 1, Exam 2, and Exam 3 have been provided to BioLINCC and dbGaP.
Supporting Information: Study Protocol, ICF
Time Frame: Data are currently available for exams 1, 2 and 3 and for cardiovascular events through 12/31/2016 and mortality through 12/31/2019. Data will be available indefinitely.
Access Criteria: Data can accessed from JHS with approved manuscript proposals and from dbGaP and BIOLINCC.
URL: https://www.jacksonheartstudy.org/

REFERENCES:
- [Background] Sempos CT, Bild DE, Manolio TA. Overview of the Jackson Heart Study: a study of cardiovascular diseases in African American men and women. Am J Med Sci. 1999 Mar;317(3):142-6. doi: 10.1097/00000441-199903000-00002. PMID 10100686
- [Background] Crook ED, Taylor H. Traditional and non-traditional risk factors for cardiovascular and renal disease in African Americans: a project of the Jackson Heart Study investigators. Am J Med Sci. 2002 Sep;324(3):115. doi: 10.1097/00000441-200209000-00001. No abstract available. PMID 12240708
- [Background] Wyatt SB, Williams DR, Calvin R, Henderson FC, Walker ER, Winters K. Racism and cardiovascular disease in African Americans. Am J Med Sci. 2003 Jun;325(6):315-31. doi: 10.1097/00000441-200306000-00003. PMID 12811228
- [Background] Crook ED, Taylor H. Traditional and nontraditional risk factors for cardiovascular and renal disease in African Americans (Part 2): a project of the Jackson Heart Study investigators. Am J Med Sci. 2003 Jun;325(6):305-6. doi: 10.1097/00000441-200306000-00001. No abstract available. PMID 12811226
- [Background] Wyatt SB, Diekelmann N, Henderson F, Andrew ME, Billingsley G, Felder SH, Fuqua S, Jackson PB. A community-driven model of research participation: the Jackson Heart Study Participant Recruitment and Retention Study. Ethn Dis. 2003 Fall;13(4):438-55. PMID 14632263
- [Background] Taylor HA Jr. Establishing a foundation for cardiovascular disease research in an African-American community--the Jackson Heart Study. Ethn Dis. 2003 Fall;13(4):411-3. PMID 14632260
- [Background] Taylor HA Jr, Clark BL, Garrison RJ, Andrew ME, Han H, Fox ER, Arnett DK, Samdarshi T, Jones DW. Relation of aortic valve sclerosis to risk of coronary heart disease in African-Americans. Am J Cardiol. 2005 Feb 1;95(3):401-4. doi: 10.1016/j.amjcard.2004.09.043. PMID 15670554
- [Background] Carpenter MA, Crow R, Steffes M, Rock W, Heilbraun J, Evans G, Skelton T, Jensen R, Sarpong D. Laboratory, reading center, and coordinating center data management methods in the Jackson Heart Study. Am J Med Sci. 2004 Sep;328(3):131-44. doi: 10.1097/00000441-200409000-00001. PMID 15367870
- [Derived] Echouffo-Tcheugui JB, Mwasongwe SE, Musani SK, Hall ME, Correa A, Hernandez AF, Golden SH, Mentz RJ, Bertoni AG. Dysglycemia and incident heart failure among blacks: The jackson heart study. Am Heart J. 2022 Mar;245:1-9. doi: 10.1016/j.ahj.2021.11.003. Epub 2021 Nov 19. PMID 34808103
- [Derived] Rao VN, Bush CG, Mongraw-Chaffin M, Hall ME, Clark D 3rd, Fudim M, Correa A, Hammill BG, O'Brien E, Min YI, Mentz RJ. Regional Adiposity and Risk of Heart Failure and Mortality: The Jackson Heart Study. J Am Heart Assoc. 2021 Jul 20;10(14):e020920. doi: 10.1161/JAHA.121.020920. Epub 2021 Jul 9. PMID 34238024
- [Derived] Rosen DM, Kundel V, Rueschman M, Kaplan R, Guo N, Wilson JG, Min YI, Redline S, Shah N. Self-reported snoring and incident cardiovascular disease events: results from the Jackson Heart Study. Sleep Breath. 2019 Sep;23(3):777-784. doi: 10.1007/s11325-018-01776-1. Epub 2019 Feb 13. PMID 30756321
- See also: Jackson Heart Study website — https://www.jacksonheartstudy.org/